CLINICAL TRIAL: NCT06320665
Title: Assessment of Vertical Pattern in Correlation With Third Molar Inclusion : a 3D CBCT Analysis
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, VANDE VANNET Bart, Professor, Central Hospital, Nancy, France
Other Study IDs: 2024PI003
Record Dates: First submitted 2024-02-06; First posted 2024-03-20 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Impacted Third Molar Tooth
Keywords: Cone beam ct; third molar; Vertical dimension; Impacted teeth; Orthodontic; Adult; Skeletal pattern
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Class I: Patient with class I occlusion, with at least one impacted third molar
  Interventions: Other: Radiographic measurement
- Class II: Patients with class II malocclusion, with at least one impacted third molar
  Interventions: Other: Radiographic measurement
- Class III: Patients with class III malocclusion, with at least one impacted third molar
  Interventions: Other: Radiographic measurement

INTERVENTIONS:
Other: Radiographic measurement — Measurements taken on 3D radiographs, to assess third molar inclusion and skeletal typology (vertical and sagittal)

SUMMARY:
The objective is to compare the sagittal and vertical skeletal parameters of patients with an impacted third molar.

Patients will be analyzed according to their skeletal characteristics: skeletal class (sagittal direction) and facial skeletal typology (vertical direction).

The inclusion characteristics of third molars will also be analyzed, to see the links between typology and inclusion. The principal hypothesis is no significant difference in third molar inclusion patterns in relation to skeletal divergence.

DETAILED DESCRIPTION:
The study is a non-interventional (observational) research involving the human person, research on existing data (retrospective study) and samples dealing with dentofacial orthopedics.

This study analyzes third molar inclusion patterns in relation with the skeletal characteristics, sagittal and vertical typology.

This is a comparative retrospective study of radiographs in three dimensions before any orthodontic treatment. The patients studied are at Bacchetti CS stage 5 (adults), and the third molar must be at least at Nolla stage 6 of formation.

There is no control group but there are subgroups depending of the skeletal characterics.

ELIGIBILITY:
Inclusion Criteria:

* CMV stage 5 on lateral radiography (end of growth)
* at least one impacted third molar at minimum Nolla stage 6 development

Exclusion Criteria:

* Previous maxillofacial trauma
* Growing patients
* Missing permanent tooth or early avulsion
* Dysplasia
* Dentofacial deformities
* Endocrinological pathologies with implications for maxillofacial growth
* Syndromes
* History of maxillofacial or orthognathic surgery
* History of orthodontic treatment
* Incomplete data

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: French adults with at least one impacted third molar
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Distance between the occlusal plane and the second molar | One day
  Depth of the third molar in mm
Angle of the third molar | One day
  The coronal-radicular axis of the mandibular third molar, and the occlusal plane of the mandibular 1st and 2nd molars, when these are in a normal, functional position on the arch (in degrees)

CONTACTS AND LOCATIONS:
Overall Officials: Bart VANDE VANNET, PhD, Study Director — Central Hospital, Nancy, France
Locations (1):
- Département d'Orthopédie dento-faciale, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Idris AM, Al-Mashraqi AA, Abidi NH, Vani NV, Elamin EI, Khubrani YH, Sh Alhazmi A, Alamir AH, Fageeh HN, Meshni AA, Mashyakhy MH, Makrami AM, Gareeb Alla Abdalla A, Jafer M. Third molar impaction in the Jazan Region: Evaluation of the prevalence and clinical presentation. Saudi Dent J. 2021 May;33(4):194-200. doi: 10.1016/j.sdentj.2020.02.004. Epub 2020 Mar 4. PMID 34025081
- [Background] Costa MG, Pazzini CA, Pantuzo MC, Jorge ML, Marques LS. Is there justification for prophylactic extraction of third molars? A systematic review. Braz Oral Res. 2013 Mar-Apr;27(2):183-8. PMID 23538430
- [Background] Hounsome J, Pilkington G, Mahon J, Boland A, Beale S, Kotas E, Renton T, Dickson R. Prophylactic removal of impacted mandibular third molars: a systematic review and economic evaluation. Health Technol Assess. 2020 Jun;24(30):1-116. doi: 10.3310/hta24300. PMID 32589125
- [Background] Tassoker M, Kok H, Sener S. Is There a Possible Association between Skeletal Face Types and Third Molar Impaction? A Retrospective Radiographic Study. Med Princ Pract. 2019;28(1):70-74. doi: 10.1159/000495005. Epub 2018 Oct 31. PMID 30380552
- [Background] Legovic M, Legovic I, Brumini G, Vandura I, Cabov T, Ovesnik M, Mestrovic S, Slaj M, Skrinjaric A. Correlation between the pattern of facial growth and the position of the mandibular third molar. J Oral Maxillofac Surg. 2008 Jun;66(6):1218-24. doi: 10.1016/j.joms.2007.12.013. PMID 18486787
- [Background] Aoun Y, Husseini B, Younes R, Ghosn N, Bouserhal J. Assessment of lower third molar space: A comparative radiographic study. Dentomaxillofac Radiol. 2022 Jul 1;51(5):20220049. doi: 10.1259/dmfr.20220049. Epub 2022 May 4. PMID 35466682
- [Background] Zamora N, Llamas JM, Cibrian R, Gandia JL, Paredes V. A study on the reproducibility of cephalometric landmarks when undertaking a three-dimensional (3D) cephalometric analysis. Med Oral Patol Oral Cir Bucal. 2012 Jul 1;17(4):e678-88. doi: 10.4317/medoral.17721. PMID 22322503
- [Background] Li C, Teixeira H, Tanna N, Zheng Z, Chen SHY, Zou M, Chung CH. The Reliability of Two- and Three-Dimensional Cephalometric Measurements: A CBCT Study. Diagnostics (Basel). 2021 Dec 7;11(12):2292. doi: 10.3390/diagnostics11122292. PMID 34943528
- [Background] Carter K, Worthington S. Predictors of Third Molar Impaction: A Systematic Review and Meta-analysis. J Dent Res. 2016 Mar;95(3):267-76. doi: 10.1177/0022034515615857. Epub 2015 Nov 11. PMID 26561441
- [Background] Bin Rubaia'an MA, Neyaz A, Talic F, Alkhamis A, Alghabban A, Assari A. The Association Between Skeletal Facial Types and Third Molars Impaction in a Saudi Arabian Subpopulation: A CBCT Study. Clin Cosmet Investig Dent. 2023 Aug 15;15:143-156. doi: 10.2147/CCIDE.S419325. eCollection 2023. PMID 37601239
- [Background] Baccetti T, Franchi L, McNamara JA Jr. An improved version of the cervical vertebral maturation (CVM) method for the assessment of mandibular growth. Angle Orthod. 2002 Aug;72(4):316-23. doi: 10.1043/0003-3219(2002)0722.0.CO;2. PMID 12169031
- [Background] Hagg U, Taranger J. Dental emergence stages and the pubertal growth spurt. Acta Odontol Scand. 1981;39(5):295-306. doi: 10.3109/00016358109162293. PMID 6950638
- [Background] Hasan KM, Sobhana CR, Rawat SK, Singh D, Mongia P, Fakhruddin A. Third molar impaction in different facial types and mandibular length: A cross-sectional study. Natl J Maxillofac Surg. 2021 Jan-Apr;12(1):83-87. doi: 10.4103/njms.NJMS_111_20. Epub 2021 Mar 16. PMID 34188406
- [Background] Mollaoglu N, Cetiner S, Gungor K. Patterns of third molar impaction in a group of volunteers in Turkey. Clin Oral Investig. 2002 Jun;6(2):109-13. doi: 10.1007/s00784-001-0144-1. PMID 12166710
- [Background] Jaron A, Trybek G. The Pattern of Mandibular Third Molar Impaction and Assessment of Surgery Difficulty: A Retrospective Study of Radiographs in East Baltic Population. Int J Environ Res Public Health. 2021 Jun 3;18(11):6016. doi: 10.3390/ijerph18116016. PMID 34205078
- [Background] Hashemipour MA, Tahmasbi-Arashlow M, Fahimi-Hanzaei F. Incidence of impacted mandibular and maxillary third molars: a radiographic study in a Southeast Iran population. Med Oral Patol Oral Cir Bucal. 2013 Jan 1;18(1):e140-5. doi: 10.4317/medoral.18028. PMID 23229243
- [Background] Ahmed M, Shaikh A, Fida M. Diagnostic validity of different cephalometric analyses for assessment of the sagittal skeletal pattern. Dental Press J Orthod. 2018 Sep-Oct;23(5):75-81. doi: 10.1590/2177-6709.23.5.075-081.oar. PMID 30427496